CLINICAL TRIAL: NCT02526056
Title: Usability and Acceptance of Exergames Among Elderly People and Physiotherapists - a Mixed Method Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Cynthia Bovard, Physiotherapist Bsc, Klinik Valens
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 15/064
Record Dates: First submitted 2015-07-09; First posted 2015-08-18 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation | interventions — Physical Therapists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapists (Experimental): The physiotherapist have to play the exergame once.
  Interventions: Other: Physiotherapists
- elderly people (Experimental): The elderly people have play the exergame twice.
  Interventions: Other: elderly people

INTERVENTIONS:
Other: Physiotherapists — This study is a usability design with qualitative and quantitative aspects. The therapeutic relevance and design features will be explored.
  Arms: Physiotherapists
Other: elderly people — In one part, with patients, physical strain and designs facets will be investigated. During their game playing process, different measurements will be done. They will be asked about their opinions about the game.
  Arms: elderly people

SUMMARY:
This study is a usability design with qualitative and quantitative aspects. In one part, with patients, physical strain and designs facets will be investigated and in another part with physiotherapists, the therapeutic relevance and design features will be explored.

For this reasons 13-15 elderly people have to play an exergame, during their game playing process, different measurements will be done. Additional 13-15 physiotherapists will also playing the exergame, they will be asked about their opinions about the game.

DETAILED DESCRIPTION:
Introduction:

The goal of a usability evaluation is to assess the degree to which a system is effective, efficient and favours positive attitudes and responses from the intended users. Exergames in particular present unique usability challenges. Because games are fundamentally different than general productivity tools, traditional usability instruments valid for productivity applications may fall short when used for serious games.

Additionally, serious games target audiences may not play games regularly; usability issues alone can hinder the game play process negatively affecting the learning experience. For this reason, user-based evaluation for exergames with adequate test user group is very important to ensure that heterogeneous population will be able to interact easily with innovative applications.

Exergames:

Exergames are defined as: ''Any number of types of video games that require the game player to physically move in order to play''.

The important aspect, in comparison to a normal videogame, is that the player uses full body movements to control on-screen action and is required to expend a significantly greater amount of energy compared with resting levels.

One of the areas that have received attention of video game researchers is that of therapeutic sessions. When exergames were used with elderly people for therapeutic sessions, it showed that special needs have to be considered.

The GameUp project:

For this reason the project GameUp was started. On their Website the project consortium state: "We will use IT technologies to promote mobility by encouraging elderly persons to be more physical active and motivating them to move more by increasing their self-efficacy". In this context exergames for elderly people were designed for Kinect® for windows. Kinect® observes all the body movements from the game player, so that they can operate the game with their body movements. In this context the game player is forced to move his body frequently in a way that increases his agility.

Therapist's view:

How do physiotherapists view the arrival of exergames in therapy rehabilitation setting, especially exergames for elderly people? Studies that focus on the therapist's view are really rare. One reference came to the conclusion that: "Video games should not be seen as a replacement of a therapist. The presence of the therapist will always be necessary for these patients to ensure that they play the game in the correct seating position, to provide mental support and social interaction during game play." But how do therapists view the use from exergames which patients could do by themselves as self-training during rehabilitation or at home? The same reference argues: "The therapist is paramount in introducing games or virtual rehabilitation to end-users; if he will not adopt the tool in his practice, neither will the patients."

Purpose of the Study:

The aim of this study is to evaluate, if elderly people accept exergames as self-training method and if this exergame is user-friendly for elderly people and physiotherapists. An additionally goal is to examine how physiotherapists evaluate the therapeutic benefit from this exergame.

Research Question:

Are exergames useable and accepted for self-training for elderly people, by themselves as well as by physiotherapists?

Design of the user trial:

This study is a usability design with qualitative and quantitative aspects. In one part, with patients, physical strain and designs facets will be investigated and in another part with physiotherapists, the therapeutic relevance and design features will be explored. Ideally the attributes required to make the product usable should be specified and measured quantitatively against predefined goals.

Number of users needed:

How many users are needed for a usability study is a controversial subject in the literature. One main point is that: "The test users should ideally reflect the serious game's target audience in terms of age, gender, education and any other demographic characteristics". In an other study is mentioned two other important aspects: It seems that serious usability problems were only found with the 13th and 15th participant. Furthermore for a usability test, it is the aim to find a study design that uncovers usability problems at the lowest cost.

In consideration of these arguments this study protocol will include 13-15 participants with different mobility levels. As the mobility level is the most important demographic character, it should be reflected by the user group.

For the physiotherapist the most important demographic character is their experience with exergames, so for this reason 13-15 physiotherapists with different experiences with exergames will be tested.

Measurements:

Heart Rate (HR):

Heart rate is an indicator of cardiovascular strain and provides an objective measure of physical work load. HR of the elderly user will be measured before playing the game, directly after finishing the game and after two minutes break.

The predefined usability criterion is: The mean HR of 80% of elderly users will be below 110 beats per minute. Previous studies have specified that heart rate between 90 and 110 indicates moderate cardiovascular strain.

Rate of Perceived Exertion (RPE):

Borg's RPE-Scale is a standardized, reliable and valid tool to describe the perception of exertion. Elderly users will be presented the Borg's 15-graded RPE scale immediately after completion of the task and will be asked to rate their perceived exertion.

The predefined usability criterion is: The RPE-score of 80% of elderly users will be below 14. This is based on previous studies where scores of more than 13 RPE have been associated with an increased relative risk for musculoskeletal symptoms.

Body Part Discomfort Scale (BPD Scale):

The Body Part Discomfort Scale has become a standard discomfort assessment tool in ergonomics research. Elderly users will be presented with a body map at the beginning and immediately after completion of the user trial.

The predefined usability criterion is: BPD Scale reports of 80% of the elderly users will be below 4. This is based on previous studies where moderate discomfort levels for any body part were selected as a threshold where redesign should be considered.

Task Analysis:

The Perceive, Recall Plan and Perform System (PRPP) is a process-oriented assessment that employs task analysis methods to determine problems with task performance. For this usability study a task analysis will be done during an elderly user or a physiotherapist is playing the game. The major task steps will be analysed to identify where the users struggles with the game design.

The predefined usability criterion for elderly user is: 80% of the elderly users can perform 60% of the needed steps without assistance.

The predefined usability criterion for the physiotherapists is: 80% of the physiotherapist can perform 80% of the needed steps without assistance.

User Questionnaire:

Furthermore to the objective measurements the users will be asked questions about their feelings and opinions about the game. Especially the physiotherapists will be asked if they see a positive therapeutic aspect and if they could imagine giving patients exergames as self-training exercises. This will be done with a questionnaire that includes open questions and five-point Likert scale questions. This is based on publications where it is considered important that the user has a positive attitude towards the product, to ensure regular and widespread use.

Data analyses:

Quantitative data will be collected to review the predefined usability criteria as specified above, using simple descriptive statistics. As sampling will be selective rather than random and the sample size will be small, statistical calculations will most likely be restricted to using median values and ranges. The median is used when no normal distribution of the data is expected and is considered a more robust value since it is not influenced by extremes.

Qualitative data will be presented as a written summary of the open questions from the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* The participants have to be older than 65 years and have had recent illness or surgery or are physiotherapists, which have a working experience at least six months with elderly patients with mobility problems.

Exclusion Criteria:

* Cognitive impairment, defined as a Mini Mental State Examination (MMSE) score < 26.
* Other disease, illness or limiting condition that would make inclusion and beneficial use of the system difficult, e.g. complete blindness or deafness or severe disabilities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change of Heart Rate | 1 day
Rate of Perceived Exertion | 1 day
Change of the Body Part Discomfort Scale | 1 day
How many percent of the needed steps are fulfilled (Task Analysis) | 1 day
  The task analysis will be done, while a Patient oder a Physiotherapist is playing the exergame. For a Task Analysis every single step, that the proband has to do is defined, e.g. press the green start button. The investigator will observe how many from the used steps the proband can do by himself. If the proband needs help, the investigator will help him and notice on which step the proband struggled.

SECONDARY OUTCOMES:
User Questionnaire | 2 day
  Acceptance and opinions about the exergame from the users (elderly people and physiotherapist),will be asked after playing the game with a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Oesch, Dr., Study Director — Kliniken Valens
Locations (1):
- Kliniken Valens, Walenstadtberg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastien JM. Usability testing: a review of some methodological and technical aspects of the method. Int J Med Inform. 2010 Apr;79(4):e18-23. doi: 10.1016/j.ijmedinf.2008.12.004. Epub 2009 Apr 2. PMID 19345139
- [Background] Wuest S, Borghese NA, Pirovano M, Mainetti R, van de Langenberg R, de Bruin ED. Usability and Effects of an Exergame-Based Balance Training Program. Games Health J. 2014 Apr 1;3(2):106-114. doi: 10.1089/g4h.2013.0093. PMID 24804155
- [Background] Plow M, Finlayson M. A qualitative study exploring the usability of Nintendo Wii Fit among persons with multiple sclerosis. Occup Ther Int. 2014 Mar;21(1):21-32. doi: 10.1002/oti.1345. Epub 2013 Apr 24. PMID 23613154
- [Background] Annema JH, Verstraete M, Abeele VV, Desmet S, Geerts D. Video games in therapy: a therapist's perspective. International Journal of Arts and Technology. 2013;6(1):106-22.
- [Background] Moreno-Ger P, Torrente J, Hsieh YG, Lester WT. Usability testing for serious games: Making informed design decisions with user data. Advances in Human-Computer Interaction. 2012;2012:4.
- [Background] GameUp. More information about GameUp. Game-Based Mobility Training and Motivation of Senior Citizens. Zaragoza (Spain): Ibernex; c2014 [cited 2015 Jan 06]. Available from: http://www.gameupproject.eu/?page_id=13. German.
- [Background] Microsoft. Meet Kinect 2015 [cited 2015 Jan 24]. Available from: http://www.microsoft.com/en-us/kinectforwindows/meetkinect/default.aspx.
- [Background] Hughes M. Rigor in Usability Testing. Technical Communication: Journal of the Society for Technical Communication. 1999;46(4):488-94.
- [Background] Åstrand P, Rodahl K. Textbook of Work Physiology: Physiological Bases of Exercise. 3 ed. Singapore: McGraw-Hill; 1986.
- [Background] Finch E, Brooks D, Strattford P, Mayo N. Physical Rehabilitation Outcome Measures. 2 ed. Hamilton: Canadian Physiotherapy Association; 2002.
- [Background] Josephson M, Hagberg M, Hjelm EW. Self-reported physical exertion in geriatric care. A risk indicator for low back symptoms? Spine (Phila Pa 1976). 1996 Dec 1;21(23):2781-5. doi: 10.1097/00007632-199612010-00014. PMID 8979326
- [Background] Corlett EN, Bishop RP. A technique for assessing postural discomfort. Ergonomics. 1976 Mar;19(2):175-82. doi: 10.1080/00140137608931530. No abstract available. PMID 1278144
- [Background] Chapparo C, Ranka J. The perceive, recall, plan, perform (PRPP) system of task analysis 2014 [cited 2015 Jan 09]. Available from: http://www.occupationalperformance.com/the-perceive-recall-plan-perform-prpp-system-of-task-analysis/.
- [Background] Faulkner X. Usability Engineering. New York 2000.
- [Background] Schädler S. Ein aufschlussreicher Test fürs Gleichgewicht. physiopraxis. 2007;5(11/12):40-1.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204